CLINICAL TRIAL: NCT06002100
Title: PREDICT: Prediction of REsponse to Depression Interventions Using Clinical and TD-fNIRS Measurements
Brief Title: Prediction of REsponse to Depression Interventions Using Clinical and TD-fNIRS Measurements
Acronym: PREDICT
Status: Enrolling by invitation | Type: Observational
Sponsor: Kernel (Industry)
Responsible Party: Sponsor
Other Study IDs: KER2023-2-PREDICT
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression; Major Depressive Disorder
Keywords: functional Near Infrared Spectroscopy (fNIRS); Ketamine; SPRAVATO; TMS; Antidepressants
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ketamine: Adult participants starting ketamine treatment for depression at a participating clinic. fNIRS measurements using Kernel Flow2 will be taken at a pre-treatment, early-treatment, and post-treatment visit. No clinical decisions will be made based on the data acquired for this study, and participation in the study has no influence on treatment decisions (including dosage form, frequency, and duration).
  Interventions: Other: fNIRS measurement
- SPRAVATO: Adult participants starting SPRAVATO treatment for depression at a participating clinic. fNIRS measurements using Kernel Flow2 will be taken at a pre-treatment, early-treatment, and post-treatment visit. No clinical decisions will be made based on the data acquired for this study, and participation in the study has no influence on treatment decisions (including dosage form, frequency, and duration).
  Interventions: Other: fNIRS measurement
- TMS: Adult participants starting TMS treatment for depression at a participating clinic. fNIRS measurements using Kernel Flow2 will be taken at a pre-treatment, early-treatment, and post-treatment visit. No clinical decisions will be made based on the data acquired for this study, and participation in the study has no influence on treatment decisions (including dosage form, frequency, and duration).
  Interventions: Other: fNIRS measurement
- Antidepressants: Adult participants starting antidepressant treatment for depression at a participating clinic. fNIRS measurements using Kernel Flow2 will be taken at a pre-treatment and short-term efficacy visit. No clinical decisions will be made based on the data acquired for this study, and participation in the study has no influence on treatment decisions (including dosage form, frequency, and duration).
  Interventions: Other: fNIRS measurement

INTERVENTIONS:
Other: fNIRS measurement — Kernel Flow2 measurements.

SUMMARY:
The purpose of the current study is to perform a unified, homogeneous data collection protocol that includes a large cohort of patients undergoing different treatment options for Major Depressive Disorder (MDD) as an avenue for investigating optimal biomarkers for depression treatments on an individual patient level.

ELIGIBILITY:
Inclusion Criteria:

Ketamine cohort

* Adult between the ages of 18 - 65, inclusive at time of enrollment
* Primary diagnosis of MDD as defined by DSM-5
* Determined by clinic to be eligible for ketamine treatment and agrees to receive ketamine treatment
* Agrees to start ketamine treatment in conjunction with study participation to capture pre-treatment measurements accurately
* Has not received a ketamine treatment course in the past 12 months
* Has not received a TMS treatment course in the past 3 months
* Ability to consent for themselves
* Fluency in English (speaking and reading)

SPRAVATO cohort

* Adult between the ages of 18 - 75, inclusive at time of enrollment
* Primary diagnosis of MDD as defined by DSM-5
* Determined by clinic to be eligible for SPRAVATO treatment and agrees to receive SPRAVATO treatment
* Agrees to start SPRAVATO treatment in conjunction with study participation to capture pre-treatment measurements accurately
* Has not received a ketamine or SPRAVATO treatment course in the past 12 months
* Has not received a TMS treatment course in the past 3 months
* Ability to consent for themselves
* Fluency in English (speaking and reading)

TMS cohort

* Adult between the ages of 18 - 65, inclusive at time of enrollment
* Primary diagnosis of MDD as defined by DSM-5
* Determined by clinic to be eligible for TMS treatment and agrees to receive TMS treatment
* Agrees to start TMS treatment in conjunction with study participation to capture pre-treatment measurements accurately
* Has not received a TMS treatment course in the past 12 months
* Has not received a ketamine or SPRAVATO treatment course within the last 3 months
* Ability to consent for themselves
* Fluency in English (speaking and reading)

Antidepressants cohort

* Adult between the ages of 18 - 65, inclusive at time of enrollment
* Primary diagnosis of MDD as defined by DSM-5
* Determined by clinic to be eligible for antidepressant treatment and agrees to receive antidepressant treatment
* Agrees to start antidepressant treatment in conjunction with study participation to capture pre-treatment measurements accurately
* Has not taken antidepressants in the past 3 months
* Has not received a TMS, SPRAVATO, or ketamine treatment course in the past 3 months
* Ability to consent for themselves
* Fluency in English (speaking and reading)

Exclusion Criteria:

* Is or may be pregnant (for participant of childbearing potential [POCBP]), even if they have been cleared to receive the depression treatment
* Unable or unwilling to wear the TD-fNIRS headset
* Has had ECT in the past 3 months
* Major visual or auditory deficits that would prevent study task completion
* Hospitalizations and/or unstable health/medical condition/treatment in the last 30 days
* Major medical illnesses and psychiatric conditions including:

  * Alzheimer's/Mild Cognitive Impairment
  * Parkinson's disease
  * Motor neuron diseases
  * Multiple Sclerosis
  * Brain Tumor
  * Stroke
  * Encephalitis
  * Meningitis
  * Epilepsy
  * TBI with serious results (coma, unconscious for >2 hrs, or skull fracture)
  * Current serious psychiatric conditions (bipolar disorder, schizophrenia, or psychosis)
* Any other clinically significant medical condition or circumstance that, in the opinion of the Investigator, could affect patient safety, preclude evaluation of response, interfere with the ability to comply with study procedures, or prohibit completion of the study
* Not an appropriate candidate for the study in the judgment of the investigator(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants seeking treatment for depression at a participating clinic/study site. Separate cohorts of participants will be enrolled depending on the treatment they have been prescribed. No clinical decisions will be made based on the data acquired for this study, and participation in the study has no influence on treatment decisions.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Brain hemodynamic activity with TD-fNIRS | Approximately 30 minutes during each study visit
  This includes changes in the concentration of oxygenated and deoxygenated hemoglobin as measured by the change in light absorption.
Optical properties of the brain with TD-fNIRS | Approximately 30 minutes during each study visit
  This measures how much light is absorbed at different points on the head.
Physiological features with TD-fNIRS | Approximately 30 minutes during each study visit
  This includes cardiac measures, such as heart rate (HR).
Physiological features with TD-fNIRS | Approximately 30 minutes during each study visit
  This includes cardiac measures, such as heart rate variability (HRV).

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | At baseline and closeout, up to 3 months
  Clinician-rated measure of depressive severity.
Patient Health Questionnaire (PHQ-9) | From baseline to closeout, up to 3 months
  9-item self-report that has been validated as a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression.
General Anxiety Disorder (GAD-7) | At baseline and closeout, up to 3 months
  7-item self-report measure used to assess participant anxiety.
Snaith-Hamilton Pleasure Scale (SHAPS) | At baseline and closeout, up to 3 months
  14-item self-administered questionnaire measuring anhedonia (inability to feel pleasure) through four domains of pleasure response: interest/pastimes, social interaction, sensory experience, and food/drink.
World Health Organization Quality of Life (WHOQOL-BREF) | At baseline and closeout, up to 3 months
  26-item self-report which aims to assess an individual's quality of life. The scale was developed with a cross-cultural approach and covers domains including physical, psychological, social relationships, and environment.
Revised Mystical Experience Questionnaire (RMEQ) | Visit 2, within approximately 7 days of baseline
  30-item self-report which provides scale scores for four domains: mystical experience, positive mood, transcendence of time and space, and ineffability. Ketamine and SPRAVATO cohorts only.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Perdue, PhD, Principal Investigator — Kernel
Locations (9):
- United States (9):
  - BrainHealth Solutions, Costa Mesa, California
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Kaizen Brain Center, LLC, La Jolla, California
  - Bespoke Treatment, Los Angeles, California
  - UCLA TMS, Los Angeles, California
  - Acacia Clinics, Sunnyvale, California
  - Metro Psychiatry Inc., Columbus, Ohio
  - Seattle Neuropsychiatric Treatment Center, Bellevue, Washington
  - Seattle Neuropsychiatric Treatment Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided